CLINICAL TRIAL: NCT07101302
Title: iCANSleep: A Randomized Controlled Trial of a Smartphone App-Based Insomnia Treatment for Cancer Survivors
Brief Title: iCANSleep: Smartphone App-Based Insomnia Treatment for Cancer Survivors
Acronym: iCANSleep
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Sheila Garland, Associate Professor of Psychology and Oncology at Memorial University of Newfoundland, Memorial University of Newfoundland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43146
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Cancer
Keywords: Cancer Survivor; Insomnia; Mobile Application
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): The immediate treatment group will begin the app-based insomnia intervention immediately after enrolling.
  Interventions: Behavioral: App-Based Cognitive Behavioural Therapy for Insomnia
- Waitlist Control (Experimental): The waitlist control group will begin the app-based intervention after a waiting period of 8 weeks after enrolling.
  Interventions: Behavioral: App-Based Cognitive Behavioural Therapy for Insomnia

INTERVENTIONS:
Behavioral: App-Based Cognitive Behavioural Therapy for Insomnia — The iCANSleep app is based on an established CBT-I protocol. The core features of the iCANSleep app include 1) a modified CBT-I protocol for cancer survivors and 2) daily sleep diaries. Core components of CBT-I treatment to be implemented include sleep restriction, stimulus control, cognitive restructuring, and psychoeducation. These components will be modified into 7-weekly modules.
  Other Names: Cognitive Behavioural Therapy for Insomnia; CBT-I

SUMMARY:
The investigators will answer the question of whether treating insomnia using the mobile-app-based intervention of Cognitive Behavioural Therapy for Insomnia (CBT-I) for cancer survivors ("iCANSleep") can improve symptoms of insomnia in Canadian cancer survivors compared to a waitlist control group. The investigators will recruit 146 people with insomnia who have completed cancer treatment at least 3 months prior to the study.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial of immediate treatment with the CBT-I app "iCANSleep" compared to a delayed treatment group with 146 cancer survivors who have completed primary treatment at least 3 months prior and meet DSM diagnostic criteria for insomnia. Participants who are randomized to the immediate treatment group will complete the 7-modules of the CBT-I treatment right away. Those randomized to the delayed treatment group will begin the intervention following an 8-week waiting period. The treatment group will complete assessments at baseline, mid-treatment, post-treatment, and 3-month follow-up. The delayed treatment group will complete an assessment at baseline, halfway through their wait at 4 weeks, and prior to beginning treatment at 8 weeks. They will also complete assessments at mid-treatment, post-treatment and 3-month follow-up. Insomnia severity will be analyzed using the Insomnia Severity Index (ISI) as the primary outcome. Other measures will include fatigue, anxiety, depression, pain, work productivity, sleep beliefs, daytime impact of insomnia, and pre-sleep arousal.

The investigators hypothesize that the immediate treatment group will report significantly greater improvements in insomnia compared to the waitlist control group at post-treatment (primary endpoint). The investigators also hypothesize that these improvements will be maintained at 3-months follow-up (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors
* Over 18 years of age
* Lives in Canada
* Understands English or French fluently
* DSM-5 diagnosis of insomnia
* ISI score of 8 or higher
* Good performance status as indicated by a score of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance status scale
* Access to internet connection
* Ownership of smartphone
* Fluency using mobile applications.
* Individuals with non-hematological malignancies must show no evidence of cancer or clinically stable/inactive disease for a minimum of 3 months prior to enrollment (for individuals with non-metastatic cancer) or be on a stable treatment regimen for the prior 3 months (for individuals with metastatic cancer) to ensure that insomnia is not a direct, acute response to cancer treatment.
* Individuals with hematological malignancies must be in remission at the time of recruitment and have completed cancer treatments (e.g., transplant, chemotherapy, immunotherapy, radiotherapy) at least 3 months prior.

Exclusion Criteria:

* Presence of a sleep disorder other than insomnia that is not adequately treated (e.g., untreated sleep apnea)
* Presence of a psychological disorder that is currently untreated or would impair the ability to participate (e.g., bipolar disorder)
* Major sensory deficit (e.g., blindness)
* Previous experience receiving CBT-I.
* The use of medications prescribed for sleep (e.g., hypnotics, sedatives, or antidepressants) will be tracked and adjusted for in the statistical analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | From enrollment until 3-month follow-up
  Insomnia Severity Index (Min: 0, Max: 28; Higher scores = worse outcomes)
Sleep Efficiency | From enrollment to end of treatment at 7 weeks
  Sleep efficiency measured by the Consensus Sleep Diary
Sleep-Onset Latency | From enrollment to end of treatment at 7 weeks
  Sleep-onset latency measured by the Consensus Sleep Diary
Wake After Sleep Onset | From enrollment to end of treatment at 7 weeks
  Wake after sleep onset measured by the Consensus Sleep Diary
Total Sleep Time | From enrollment to end of treatment at 7 weeks
  Total sleep time measured by the Consensys Sleep Diary

SECONDARY OUTCOMES:
Fatigue | From enrollment to 3-month follow-up
  Patient-Reported Outcome Measurement Information System: Fatigue 8a Short Form (Min: 8, Max: 40; Higher scores = worse outcomes)
Anxiety | From enrollment to 3-month follow-up
  Patient-Reported Outcome Measurement Information System Anxiety 8a Short Form (Min: 8, Max: 40; Higher scores = worse outcomes)
Depression | From enrollment to 3-month follow-up
  Patient-Reported Outcome Measurement Information System Depression 8a Short Form (Min: 8, Max: 40; Higher scores = worse outcomes)
Pain Level | From enrollment to 3-month follow-up
  Patient-Reported Outcome Measurement Information System Pain 8a Short Form (Min: 8, Max: 40; Higher scores = worse outcomes)
Cognitive Function | From enrollment to 3-month follow-up
  Patient-Reported Outcome Measurement Information System Cognitive Function 8a Short Form (Min: 8, Max: 40; Higher scores = worse outcomes)
Work Productivity and Activity Impairment | From enrollment to 3-month follow-up
  Work Productivity and Activity Impairment (WPAI; Min: 0%, Max: 100%; Higher scores = greater impairment)
App Engagement | From time of starting the app to completing treatment (7 weeks)
  App engagement will be measured based on the number of logins, complete session use (duration of time on the app), number of visits and amount of time on each module, use of the daily sleep journal and engagement with extra resources and support material.
Adverse Events | From enrollment to 3-month follow-up
  There is no validated method of reporting AEs in trials of CBT-I in cancer populations. As such, we will use the method developed for the Addressing Cancer Treatment-Related Insomnia Online in Atlantic Canada (ACTION) study, based on the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 and the National Cancer Institute, Cancer Therapy Evaluation Program attribution standards. AEs will be assessed using open- and closed-ended questions. This method follows the CONSORT 2022 guidelines for reporting harms to ensure that the: (1) AEs are clearly defined with descriptions of anticipated AEs; (2) Measurement of AEs and methodology are clearly stated, including validation of measures and timing of use; (3) AEs are reported with an attribution to the relationship of the intervention (i.e. is the AE actually related to the intervention?); and (4) Severity of each AE is reported. This measure will be administered at mid-treatment (4 weeks) and post-treatment (8 weeks).
Sleep-Related Beliefs | From enrollment to 3-month follow-up
  Cancer-related dysfunctional beliefs and attitudes about sleep (C-DBAS-14; Min: 0, Max: 140; Higher scores = more dysfunctional beliefs)
Pre-Sleep Arousal | From enrollment to 3-month follow-up
  Pre-sleep arousal scae (PSAS; Min: 16, Max: 80; Higher scores = worse outcomes)
Sleep Metrics | During 8-week waiting period for waitlist control group and from treatment end (7 weeks) to 3-month follow up
  Whole week Self Assessment of sleep survey (SASS)
Daytime Impact of Insomnia | From enrollment to 3-month follow-up
  Insomnia daytime symptom and impact questionnaire (IDSIQ; Min: 0, Max: 140; Higher scores = worse outcomes)
Smartphone Self-Efficacy | Baseline
  The Smartphone Self-Efficacy Scale (SSES; Min: 19, Max: 95; Higher scores = worse outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila N Garland, Principal Investigator — Memorial University of Newfoundland; Rachel M Lee, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The official iCANSleep study website — https://icansleep.app